CLINICAL TRIAL: NCT00040001
Title: Safety and Efficacy Study of an A1-Adenosine Receptor Agonist to Slow Heart Rate in Atrial Fibrillation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aderis Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DTI-0009/003
Record Dates: First submitted 2002-06-18; First posted 2002-06-20 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — selodenoson

INTERVENTIONS:
Drug: DTI-0009

SUMMARY:
This study is designed to evaluate the safety of DTI-0009 in patients with atrial fibrillation and to find the dose of DTI-0009 that lowers heart rates in patients with atrial fibrillation with rapid ventricular response.

ELIGIBILITY:
Inclusion Criteria

* Primary diagnosis of atrial fibrillation with rapid ventricular response of any duration as documented by an ECG

Exclusion Criteria

* Presence of other significant cardiac disease or history of significant neurological, hepatic,cardiovascular, renal, gastrointestinal, thyroid, respiratory, rheumatologic, or hematologic disease or impairment that in the investigator's judgment is serious enough to preclude the patient from safely participating in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple locations, Richmond, Virginia, United States